CLINICAL TRIAL: NCT04539106
Title: Clinical Outcome Following Reinjection of Ranibizumab in Recurrent Cases With Retinopathy of Prematurity
Brief Title: Intravitreal Ranibizumab in Recurrent ROP
Status: Completed | Type: Observational
Sponsor: Ameera Gamal Abdelhameed (Other)
Responsible Party: Sponsor-Investigator, Ameera Gamal Abdelhameed, Lecturer of Ophthalmology, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: intravitreal Ranibizumab reinj
Record Dates: First submitted 2020-08-26; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: intravitreal injection of Ranibizumab — intravitreal injection of 0.25 mg/0.025 ml ranibizumab with a 30-gauge needle 1.5mm from limbus

SUMMARY:
A retrospective study included reviewing of medical records of preterm babies who were admitted in neonatal intensive care unit (NICU) of Mansoura University children hospital (MUCH) or referred from nearby hospitals for ROP screening during the period from March 2013 to February 2020.

DETAILED DESCRIPTION:
Retinopathy of prematurity was diagnosed and classified according to the International Classification of ROP. Data of the patients who received IVR for type 1 ROP or aggressive posterior ROP (AP-ROP) according to early treatment ROP study (ETROP) were collected. Intravitreal ranibizumab injection was performed as follows; topical anesthetic drop was applied, standard aseptic eye preparation with 5% betadine was performed, a lid speculum was inserted and intravitreal injection of 0.25 mg/0.025 ml ranibizumab with a 30-gauge needle 1.5mm from limbus was given. In case of bilateral ROP, both eyes are injected in the same session. Infants were examined a day after the procedure and weekly thereafter until full vascularization of the retina was observed.

ROP reactivation was defined as any of the following: recurrent plus disease, recurrent neovascularization, or reformation of ridge despite treatment . Once recurrence was determined, second injection of IVR (0.25mg/0.025mL) was given to patients or surgery was performed if progressed to stage 4 or 5. All treated infants were examined until complete regression of ROP and full retinal vascularization.

ELIGIBILITY:
Inclusion Criteria:

* patients received IVR for type 1 ROP or aggressive posterior ROP (AP-ROP) according to early treatment ROP study (ETROP) and developed recurrence of ROP

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ROP reactivation was defined as any of the following: recurrent plus disease, recurrent neovascularization, or reformation of ridge despite treatment
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
full vascularization of the retina | 6 months
  Infants were examined a day after the procedure and weekly thereafter until full vascularization of the retina was observed.

CONTACTS AND LOCATIONS:
Overall Officials: Rania MR Bassiouny, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Lad EM, Hernandez-Boussard T, Morton JM, Moshfeghi DM. Incidence of retinopathy of prematurity in the United States: 1997 through 2005. Am J Ophthalmol. 2009 Sep;148(3):451-8. doi: 10.1016/j.ajo.2009.04.018. Epub 2009 Jul 9. PMID 19541285
- [Background] Gilbert C. Retinopathy of prematurity: a global perspective of the epidemics, population of babies at risk and implications for control. Early Hum Dev. 2008 Feb;84(2):77-82. doi: 10.1016/j.earlhumdev.2007.11.009. Epub 2008 Jan 29. PMID 18234457
- [Background] Kwinta P, Bik-Multanowski M, Mitkowska Z, Tomasik T, Pietrzyk JJ. The clinical role of vascular endothelial growth factor (VEGF) system in the pathogenesis of retinopathy of prematurity. Graefes Arch Clin Exp Ophthalmol. 2008 Oct;246(10):1467-75. doi: 10.1007/s00417-008-0865-9. Epub 2008 Jun 11. PMID 18546007
- [Background] Multicenter trial of cryotherapy for retinopathy of prematurity. Preliminary results. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1988 Apr;106(4):471-9. doi: 10.1001/archopht.1988.01060130517027. PMID 2895630
- [Background] McNamara JA, Tasman W, Brown GC, Federman JL. Laser photocoagulation for stage 3+ retinopathy of prematurity. Ophthalmology. 1991 May;98(5):576-80. doi: 10.1016/s0161-6420(91)32247-4. PMID 2062488
- [Background] Hunter DG, Repka MX. Diode laser photocoagulation for threshold retinopathy of prematurity. A randomized study. Ophthalmology. 1993 Feb;100(2):238-44. doi: 10.1016/s0161-6420(93)31664-7. PMID 8437833
- [Background] Iverson DA, Trese MT, Orgel IK, Williams GA. Laser photocoagulation for threshold retinopathy of prematurity. Arch Ophthalmol. 1991 Oct;109(10):1342-3. doi: 10.1001/archopht.1991.01080100022007. No abstract available. PMID 1929909
- [Background] Mintz-Hittner HA, Kennedy KA, Chuang AZ; BEAT-ROP Cooperative Group. Efficacy of intravitreal bevacizumab for stage 3+ retinopathy of prematurity. N Engl J Med. 2011 Feb 17;364(7):603-15. doi: 10.1056/NEJMoa1007374. PMID 21323540
- [Background] Lin CJ, Chen SN, Tseng CC, Chang YC, Hwang JF. Effects of ranibizumab on very low birth weight infants with stage 3 retinopathy of prematurity: A preliminary report. Taiwan Journal of Ophthalmology 2012; 2: 136-139
- [Background] Bakri SJ, Snyder MR, Reid JM, Pulido JS, Ezzat MK, Singh RJ. Pharmacokinetics of intravitreal ranibizumab (Lucentis). Ophthalmology. 2007 Dec;114(12):2179-82. doi: 10.1016/j.ophtha.2007.09.012. PMID 18054637
- [Background] Krohne TU, Liu Z, Holz FG, Meyer CH. Intraocular pharmacokinetics of ranibizumab following a single intravitreal injection in humans. Am J Ophthalmol. 2012 Oct;154(4):682-686.e2. doi: 10.1016/j.ajo.2012.03.047. Epub 2012 Jul 19. PMID 22818800
- [Background] Bakri SJ, Snyder MR, Reid JM, Pulido JS, Singh RJ. Pharmacokinetics of intravitreal bevacizumab (Avastin). Ophthalmology. 2007 May;114(5):855-9. doi: 10.1016/j.ophtha.2007.01.017. PMID 17467524
- [Background] Mireskandari K, Adams GG, Tehrani NN. Recurrence of retinopathy of prematurity following bevacizumab monotherapy: is it only the tip of the iceberg? JAMA Ophthalmol. 2013 Apr;131(4):544-5. doi: 10.1001/jamaophthalmol.2013.711. No abstract available. PMID 23579608